CLINICAL TRIAL: NCT04139707
Title: An Information and Computer Technology-based Mobile Application for Training of Family Members Caring for Someone With Dementia
Brief Title: A Mobile Application for Training of Family Caregivers Caring for Someone With Dementia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Amine Choukou, Assistant Professor, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HS23111 (H2019:319)
Record Dates: First submitted 2019-10-21; First posted 2019-10-25 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Dementia
Keywords: dementia; care-giving; communication; mobile application
MeSH Terms: conditions — Dementia; Communication

STUDY DESIGN:
Intervention Model Description: Pilot Randomized Controlled Trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Caring4Dementia Group (Experimental): The experimental group will receive Careing4Dementia downloadable on their smartphone or tablet. Caring4Dementia will tell and show caregivers of a person living with dementia how to 1) manage difficult behaviors, 2) deal with refusal, 3) deal with tensions and 4) manage work-life demands. The app is self-administered and self-paced and contains surveys referring to the outcome measurements tools used in the study. The intervention will be for 30 days without any restriction or limitation in terms of timing, location or frequency of use.
  Interventions: Device: Caring4Dementia
- White Paper Group (Active Comparator): The White Paper group will receive a white paper on the principles of communicating efficiently with persons living with dementia.
  Interventions: Other: White Paper
- Control Goup (No Intervention): The control group will not receive any intervention.

INTERVENTIONS:
Device: Caring4Dementia — A mobile application administered for 30 days, which provides people caring for a person living with dementia with a useful and intuitive tool targeting communication skills.
  Arms: Caring4Dementia Group
Other: White Paper — The White Paper group will receive a white paper (hard copy and electronically) on the principles of communicating efficiently with persons living with dementia.
  Arms: White Paper Group

SUMMARY:
Background

The mental, physical, and emotional health of caregivers is negatively affected by the burden of caring for of persons living with dementia. Caregivers are usually reported as feeling frustrated, angry, exhausted, guilty, helpless and unable to bear the heavy burden of their caregiving responsibilities. In addition to depressive symptoms and other mental health problems among caregivers, the physical stress of caring for someone who is unable to perform daily activities such as bathing, grooming and other personal care, has been shown to be a serious threat to caregivers' physical health outcomes. Evidence has shown that greater levels of stress, anxiety, depression, frustration, and lower subjective well-being and self-efficacy are exhibited in a greater amount among family and friends who care for persons living with dementia compared to those who do not have the burden of caring for a persons living with dementia. Caregivers have been shown to use alcohol and other drugs at a higher rate than those who do not need to care for others as a reaction to this increased stress. Studies has also shown that caregivers are more likely than non-Caregivers to use opioid or psychotropic medications. One over five caregivers (22%) feel tired when they go to bed at night.

Objectives

This study relies on a mobile application (Caring4Dementia) that provides people, caring for a person living with dementia, with a useful and intuitive training tool targeting communication skills. The aims of this study are to evaluate the feasibility and acceptability of using Caring4Dementia within a self-administered program and the preliminary efficacy of the Caring4Dementia intervention.

ELIGIBILITY:
Inclusion Criteria:

* Informal caregiver of a person living with dementia for more than 6 months
* Able to read and understand English
* Able to use smartphones and tablets (Apple or Android)
* Have a smartphone or tablet (Apple or Android) with internet connection, involved in this study
* 18 years or over
* Give written and oral informed consent

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-01-02 (Actual); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in caregiver well-being | Baseline (Day 1), post (day 30), Retention (90 days) after baseline
  Measured by the Caregiver Well-Being Scale to determine the frequency in which basic needs and activities of living have been met for the caregiver within the last three months. Items in this self-reported scale are scored on a 5-point scale [ranging form "Rarely (1)" to "Usually (5)"], with a higher dimension score indicating greater intensity in that dimension. The highest score possible is 70, meaning a higher well-being.

SECONDARY OUTCOMES:
Change in caregiver burden | Baseline (Day 1), post (day 30), Retention (90 days) after baseline
  Measured by the Short version of the Burden Scale for Family Caregivers. This is a 10-item instrument. Each item is a statement that is rated on a 4-point scale with the values "strongly disagree" (0), "disagree" (1), "agree" (2), and "strongly agree" (3). The scale ranges from 0 to 30, with a higher dimension score indicating greater intensity in that dimension.
Change in caregivers' perceived challenges and resources | Baseline (Day 1), post (day 30), Retention (90 days) after baseline
  Measured by the Adult Carer Quality of Life Questionnaire, a 40-item instrument that measures the overall quality of life for adult carers, and subscale scores for eight domains of quality of life. Scores on the overall questionnaire have a possible range of 0 to 120 with higher scores indicating greater quality of life.
Activity volume on the Caring4Dementia app | 30 days
  Usage logs will be saved on the cloud to quantify the time (s) spent on every activity for all the activities.
Activity frequency on the Caring4Dementia app | 30 days
  Usage logs will be saved on the cloud to quantify the frequency of use of every activity in the application for all the activities (how many time per day the caregiver engage in the activity).

CONTACTS AND LOCATIONS:
Locations (1):
- Riverview Health Centre, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No